CLINICAL TRIAL: NCT05841017
Title: Effectiveness of the Immersive Virtual Reality in the Psychological Treatment of Obsessive Compulsive Disorder
Brief Title: Immersive Virtual Reality & Obsessive Compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Consorci Hospitalari de Vic (Other)
Responsible Party: Principal Investigator, Dr. Pere Roura-Poch, Head of Epidemiology, Consorci Hospitalari de Vic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-282
Record Dates: First submitted 2023-03-29; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Immersive Virtual Reality; psychological treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will participate in a psychoeducational group (1) and in individual psychological intervention based in Cognitive Behavioural Therapy (2).
  Interventions: Behavioral: Psychotherapy with Immersive Virtual Reality support.
- Control group (No Intervention): Usual clinic care.

INTERVENTIONS:
Behavioral: Psychotherapy with Immersive Virtual Reality support. — Psychoeducational group intervention and cognitive behavioural therapy individual intervention.
  Arms: Intervention group

SUMMARY:
Immersive VR (IVR) is based on the generation and projection of images from different perspectives. Obsessive Compulsive Disorder (OCD) is considered one of the 5 most common mental disorders and one of the 20 most disabling diseases according to the World Health Organization (WHO). Its vital prevalence is about 2.5%. This study aims to establish the effectiveness of a cognitive-behavioral intervention - individual and group - using IVR in patients diagnosed with OCD compared to a group receiving standard treatment by the Mental Health Center. A sample will be obtained from the list of all patients registered in the Mental Health Service of the University Hospital of Vic (Vic, Catalonia) with the primary or secondary diagnosis of Obsessive Compulsive Disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM 5) and in active treatment status in the period between January 2021 and January 2023. Randomized controlled clinical trial. Variables: sociodemographic, clinical, OCD symptom follow-up and quality of life. Measurement instruments: Yale-Brown Obsessive Compulsive Scale (Y-BOCS), State-Trait Anxiety Inventory (STAI), Beck Depression Inventory (BDI), Immersive Tendencies Questionnaire (ITQ), Presence Questionnaire, EuroQoL-5D (EQ-5D). Inclusion criteria: Patients over 18 years of age with a primary or secondary diagnosis of Obsessive Compulsive Disorder with one of the following specifiers: with good or acceptable introspection (1) or with little introspection (2); persons with current activity at the Mental Health Center. Exclusion criteria: patients with a diagnosis of intellectual disability, autistic spectrum disorder, active substance-related disorders, neuro-cognitive disorder and/or severe personality disorder; acute psychopathological decompensation; insufficient command of Catalan and/or Spanish; advanced disease and/or disease that significantly hinders the follow-up of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age)
* Outpatient
* Current diagnostic of obsessive compulsive disorder with good or fair insight (1) or with poor insight (2)
* Follow-up by mental health network in Vic Hospital Consortium of Catalonia
* Signed informed consent

Exclusion Criteria:

* Intellectual disabilities
* Autism spectrum disorder
* Active substance-related disorders
* Neurocognitive disorders
* Several personality disorders
* Clinical acute psychotic relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-08-11 (Estimated); Study Completion 2024-02-12 (Estimated)

PRIMARY OUTCOMES:
Obsessive Compulsive Disorder symptomatology. | 1, 3 & 6 months.
  Changes in score of Yale-Brown Obsessive Compulsive Scale (Y-BOCS). Total score 0-40. Subclinical level (0-7); mild (8-15); moderate (16-23); severe (24-31) and very severe (32-40). Changes in minor categories and reduction in scores indicate improvement.

SECONDARY OUTCOMES:
Anxiety symptoms. | 1, 3 & 6 months.
  Changes in score of State-Trait Anxiety Inventory (STAI). Total score of State Anxiety and in Trait Anxiety is between 0-60. Decreased scores indicate improvement.
Depressive mood symptoms. | 1, 3 & 6 months.
  Changes in score of Beck Depression Inventory (BDI). Score range 0-63. The scores obtained would indicate low depression (0-13); mild depression (14-19); moderate depression (20-28) and severe depression (29-63). Changes in minor categories and reduction in scores indicate improvement.
Perceived quality of life. | 1, 3 & 6 months.
  Changes in score of European Quality of Life - 5 Dimensions (EuroQoL-5D). This scale consists of two parts, a first part that evaluates 5 dimensions: mobility, personal care, daily activities, pain/discomfort and anxiety/depression. The second part consists of a visual analogue scale graduated from 0 (worst imaginable state of health) to 100 (best imaginable state of health). In first part, lower score indicate better outcomes. In last part, higher score indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Roura-Poch, MD, Study Chair — Consorci Hospitalari de Vic
Locations (1):
- Consorci Hospitalari de Vic, Vic, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fineberg NA, Hollander E, Pallanti S, Walitza S, Grunblatt E, Dell'Osso BM, Albert U, Geller DA, Brakoulias V, Janardhan Reddy YC, Arumugham SS, Shavitt RG, Drummond L, Grancini B, De Carlo V, Cinosi E, Chamberlain SR, Ioannidis K, Rodriguez CI, Garg K, Castle D, Van Ameringen M, Stein DJ, Carmi L, Zohar J, Menchon JM. Clinical advances in obsessive-compulsive disorder: a position statement by the International College of Obsessive-Compulsive Spectrum Disorders. Int Clin Psychopharmacol. 2020 Jul;35(4):173-193. doi: 10.1097/YIC.0000000000000314. PMID 32433254
- [Background] Hamatani S, Tsuchiyagaito A, Nihei M, Hayashi Y, Yoshida T, Takahashi J, Okawa S, Arai H, Nagaoka M, Matsumoto K, Shimizu E, Hirano Y. Predictors of response to exposure and response prevention-based cognitive behavioral therapy for obsessive-compulsive disorder. BMC Psychiatry. 2020 Sep 4;20(1):433. doi: 10.1186/s12888-020-02841-4. PMID 32887553
- [Background] Laforest M, Bouchard S, Bosse J, Mesly O. Effectiveness of In Virtuo Exposure and Response Prevention Treatment Using Cognitive-Behavioral Therapy for Obsessive-Compulsive Disorder: A Study Based on a Single-Case Study Protocol. Front Psychiatry. 2016 Jun 13;7:99. doi: 10.3389/fpsyt.2016.00099. eCollection 2016. PMID 27378951
- [Background] Langener S, Van Der Nagel J, van Manen J, Markus W, Dijkstra B, De Fuentes-Merillas L, Klaassen R, Heitmann J, Heylen D, Schellekens A. Clinical Relevance of Immersive Virtual Reality in the Assessment and Treatment of Addictive Disorders: A Systematic Review and Future Perspective. J Clin Med. 2021 Aug 18;10(16):3658. doi: 10.3390/jcm10163658. PMID 34441953
- [Background] van Bennekom MJ, de Koning PP, Gevonden MJ, Kasanmoentalib MS, Denys D. A Virtual Reality Game to Assess OCD Symptoms. Front Psychiatry. 2021 Jan 22;11:550165. doi: 10.3389/fpsyt.2020.550165. eCollection 2020. PMID 33551856